CLINICAL TRIAL: NCT00167180
Title: Use of Cyclophosphamide/Fludarabine to Promote in Vivo Expansion of Donor Lymphocyte Infusions (DLI) to Enhance Efficacy After Allogeneic Transplant
Brief Title: Post Transplant Donor Lymphocyte Infusion
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Accrual Goal Met
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004LS006; MT2003-15 (Other: Blood and Marrow Transplantation Program); 0401M55207 (Other: IRB, University of Minnesota); NCT00303693 (obsolete NCT alias)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Leukemia, Myeloid, Chronic; Lymphomas; Multiple Myeloma; Myelodysplastic Syndrome; Leukemia, Lymphocytic, Acute; Leukemia, Lymphocytic, Chronic; AML
Keywords: donor lymphocyte infusions; BMT; bone marrow transplant
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Lymphoma; Multiple Myeloma; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Induction Chemotherapy; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CML (Active Comparator): Patients with Chronic Myelogenous Leukemia (CML) who have failed or refused Gleevec(TM) therapy and will receive Donor Lymphocyte Infusion.
  Interventions: Procedure: Donor Lymphocyte Infusion
- Non-CML or CML that Relapsed after Donor Lymphocyte Infusion (Active Comparator): Patients with non-CML or CML who have failed Donor Lymphocyte Infusion (DLI) and will receive induction chemotherapy plus DLI.
  Interventions: Procedure: Donor Lymphocyte Infusion; Drug: Induction Chemotherapy

INTERVENTIONS:
Procedure: Donor Lymphocyte Infusion — donor cells infused over 2 hrs at cell dose of 0.5 dx 10^8 CD3+T-cells/kg
  Other Names: DLI
Drug: Induction Chemotherapy — Fludarabine 25 mg/m2 IV Cyclosphosphamide 60 mg/kg IV
  Other Names: Fludara; Endoxan, Cytoxan, Neosar, Procytox, Revimmune, cytophosphane
  Arms: Non-CML or CML that Relapsed after Donor Lymphocyte Infusion

SUMMARY:
The purpose of this study is to test the hypothesis that a pre-infusion preparative regimen of cyclophosphamide and fludarabine will improve the effectiveness of DLI in patients with blood cancers.

DETAILED DESCRIPTION:
When cancer relapses after donor bone marrow transplantation, regular dose chemotherapy offers little hope of prolonged survival. However, there is evidence that lymphocytes can attack cancer cells. There is considerable evidence that this immune attack on cancer cells is associated with graft-versus-host disease. Although graft-versus-host disease can cause problems, this immune reaction may, in part, be the way that bone marrow transplantation cures cancer. In this study we hope that infusion of immune cells from the subject's bone marrow donor plus a chemotherapy regimen of cyclophosphamide and fludarabine will activate the subject's immune system to attack their cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients (age > or = 1 years) with a diagnosis of relapse after related or unrelated allogeneic stem cell transplantation for a hematological malignancy.
* For CML, relapse will be defined as any cytogenetic evidence of a Philadelphia chromosome or persistence of BCR/ABL rearrangements by molecular testing on at least two measurements over a 6 month interval. If cytogenetics are normal and there is PCR evidence of a BCR/ABL fusion, patients will be eligible if they have evidence of a quantitative increase in CML measured either by quantitative PCR or by fluorescent in situ hybridization (FISH).
* For non-CML, relapse will be defined based on disease specific morphologic criteria from a bone marrow biopsy and aspirate or recurrence of disease specific cytogenetics. For disease specific definition of relapse, see appendix 3. Relapse can be determined morphologically with less than 5 percent blasts if definitive relapse can be determined. Equivocal results for relapse should result in a repeated test after an appropriate time interval (suggested 1 month) to determine eligibility.

Post-transplant lymphoproliferative diseases (often referred to as EBV-associated lymphomas) are NOT eligible for this protocol.

* For Chronic Phase CML patients only
* - must have failed (no response in 3 months or incomplete response at 6 months) or refused treatment with Gleevec
* - if no prior DLI, CML patients will first have DLI- if relapse occurs after DLI, DLI with chemotherapy per this protocol will be offered
* Patients must be within one year of identification of relapse or if beyond that time period, must have at least 10% donor DNA by RFLP or cytogenetics.
* Same allogeneic donor (sibling or URD) used for transplantation is available for lymphocyte donation.
* No severe organ damage (by laboratory or clinical assessment) as measured by:
* - blood creatinine ≤ 2.0 mg/dL
* - liver function tests < 5 x normal
* - left ventricular ejection fraction > 40% (testing required only if symptomatic or prior known impairment).
* - pulmonary functions > 50% (testing required only if symptomatic or prior known impairment). Oxygen saturation (>92%) can be used in child where PFT's cannot be obtained.
* - chest x-ray without evidence of active infection
* Off prednisone and other immunosuppressive agents (given for any reason) for at least 3 days prior to DLI infusions.
* Performance status ≥ 60%
* Women must not be pregnant or lactating. The agents used in this study may be teratogenic to a fetus and there is no information on the excretion of agents into breast milk All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy
* Women of childbearing potential and sexually active males are strongly advised to use an accepted and effective method of contraception
* Patient must given written informed consent indicating understanding of the nature of the treatment and its potential risks

Exclusion Criteria:

* Concurrent signs of acute or chronic graft-versus-host disease requiring ongoing treatment at the time of relapse will be ineligible.
* Patients being treated for GVHD with prednisone, cyclosporine, Imuran or other immunosuppressive medications are not eligible until these medications are discontinued for at least 2 weeks without a flare of GVHD.
* Active CNS leukemia
* Active fungal infection or pulmonary infiltrates (stable prior treated disease is allowable)
* HIV positive

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2004-01; Primary Completion 2017-11-21 (Actual); Study Completion 2018-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Miller, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Miller JS, Weisdorf DJ, Burns LJ, Slungaard A, Wagner JE, Verneris MR, Cooley S, Wangen R, Fautsch SK, Nicklow R, Defor T, Blazar BR. Lymphodepletion followed by donor lymphocyte infusion (DLI) causes significantly more acute graft-versus-host disease than DLI alone. Blood. 2007 Oct 1;110(7):2761-3. doi: 10.1182/blood-2007-05-090340. Epub 2007 Jun 19. PMID 17579184

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the recruitment period of the study, the donor lymphocyte infusion (DLI) was reduced from 1.0 x 10^8 CD3+ T-cells/kg to 0.5 x 10^8 CD3+ T-cells/kg due to an excess rate and intensity of graft vs. host disease.
Groups:
- Chronic Myelogenous Leukemia (CML): Patients who have failed or refused Gleevec (TM) therapy and will receive Donor Lymphocyte Infusion.
  Donor Lymphocyte Infusion: donor cells infused over 2 hrs at cell dose of 0.5 dx 10^8 CD3+T-cells/kg
- Non-CML or CML Failing Donor Lymphocyte Infusion: Patients with non-CML or CML who have failed DLI and will receive Induction Chemotherapy + DLI.
  Induction Chemotherapy + DLI: Fludarabine 25 mg/m2 IV Cyclosphosphamide 60 mg/kg IV Donor Lymphocyte Infusion (DLI)
Period: Overall Study
Arm/Group | Chronic Myelogenous Leukemia (CML) | Non-CML or CML Failing Donor Lymphocyte Infusion
Started | 0 | 57
Completed | 0 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- DLI Cell Dose of 1.0 x 10^8 CD3+ T-cells/kg: Cyclophosphamide 60mg/kg IV over 2 hours Fludarabine 25 mg/m2 IV over 30 minutes DLI Cell Dose 1.0 x 10^8 CD3+ T-cells/kg
- DLI Cell Dose of 0.5 x 10^8 CD3+ T-cells/kg: Cyclophosphamide 60mg/kg IV over 2 hours Fludarabine 25 mg/m2 DLI Cell Dose 0.5 x 10^8 CD3+ T-cells/kg
- Total: Total of all reporting groups
Arm/Group | DLI Cell Dose of 1.0 x 10^8 CD3+ T-cells/kg | DLI Cell Dose of 0.5 x 10^8 CD3+ T-cells/kg | Total
Number analyzed (Participants) | 15 | 42 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 14 | 36 | 50
  >=65 years | 0 | 4 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 18 | 25
  Male | 8 | 24 | 32
Race (NIH/OMB) [Count of Participants; unit: Participants] — Due to this study starting about 15 years ago, this data is not accessible at this point. The race data WAS collected, but it was collected on all of the patients, but was not split by arm so there is not way at this point to separate the demographic data by arm. If it's possible to report the race data on the trial as a whole instead of by arm, please let me know! As of now, I have entered this in as accurate as possible given the data available to me.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 3 | 3
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 1 | 1
    White | 15 | 38 | 53
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Alive
Description: The percentage of people in a study or treatment group who are alive for a certain period of time after they were diagnosed with or treated for a disease, such as cancer. Also called survival rate.
  Overall survival will be defined as time from date of enrollment to date of death or censored at the date of last documented contact for patients still alive.
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | DLI Cell Dose of 1.0 x 10^8 CD3+ T-cells/kg | DLI Cell Dose of 0.5 x 10^8 CD3+ T-cells/kg
Number analyzed (Participants) | 15 | 42
Participants | 3 | 20

2. Secondary Outcome: Number of Patients Alive Without Disease
Description: The number of patients alive one year after treatment without any signs or symptoms of the cancer being treated or any other type of cancer. In a clinical trial, measuring the disease-free survival is one way to see how well a new treatment works.
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | DLI Cell Dose of 1.0 x 10^8 CD3+ T-cells/kg | DLI Cell Dose of 0.5 x 10^8 CD3+ T-cells/kg
Number analyzed (Participants) | 15 | 42
Participants | 2 | 10

3. Secondary Outcome: Number of Participants With Complete Remission
Description: In complete remission, all signs and symptoms of cancer that can be detected with modern technology have disappeared, although cancer still may be in the body.
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | DLI Cell Dose of 1.0 x 10^8 CD3+ T-cells/kg | DLI Cell Dose of 0.5 x 10^8 CD3+ T-cells/kg
Number analyzed (Participants) | 15 | 42
Participants | 7 | 22

4. Secondary Outcome: Number of Patients With Acute Graft-Versus-Host Disease
Description: Acute Graft-Versus-Host Disease is a severe short-term complication created by infusion of donor cells into a foreign host.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | DLI Cell Dose of 1.0 x 10^8 CD3+ T-cells/kg | DLI Cell Dose of 0.5 x 10^8 CD3+ T-cells/kg
Number analyzed (Participants) | 15 | 42
Participants | 10 | 10

5. Secondary Outcome: Number of Patients With Bone Marrow Aplasia
Description: Aplastic anemia is a disorder in which the bone marrow greatly decreases or stops production of blood cells.
  In aplastic anemia, the basic structure of the marrow becomes abnormal, and those cells responsible for generating blood cells (hematopoietic cells) are greatly decreased in number or absent. These hematopoietic cells are replaced by large quantities of fat.
Time Frame: Day 100
Measure: Count of Participants; unit: Participants
Arm/Group | DLI Cell Dose of 1.0 x 10^8 CD3+ T-cells/kg | DLI Cell Dose of 0.5 x 10^8 CD3+ T-cells/kg
Number analyzed (Participants) | 15 | 42
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | DLI Cell Dose of 1.0 x 10^8 CD3+ T-cells/kg | DLI Cell Dose of 0.5 x 10^8 CD3+ T-cells/kg
All-Cause Mortality (participants affected / at risk) | 12/15 | 22/42
Serious Adverse Events (participants affected / at risk) | 8/15 | 3/42
Other Adverse Events (participants affected / at risk) | 12/15 | 11/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DLI Cell Dose of 1.0 x 10^8 CD3+ T-cells/kg (N=15) | DLI Cell Dose of 0.5 x 10^8 CD3+ T-cells/kg (N=42)
Death, NOS (General disorders) | 1 | 0
Acute Graft vs. Host Disease (General disorders) | 7 | 1
Infection, NOS (Infections and infestations) | 1 | 0
Acute Sepsis (Infections and infestations) | 1 | 0
Pulmonary Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Graft vs. Host Disease, NOS (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DLI Cell Dose of 1.0 x 10^8 CD3+ T-cells/kg (N=15) | DLI Cell Dose of 0.5 x 10^8 CD3+ T-cells/kg (N=42)
Acute Graft vs. Host Disease (General disorders) | 6 | 0
Acute Renal Failure (Renal and urinary disorders) | 0 | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaphylactic Reaction to Anti-Thymocyte Globulin (Immune system disorders) | 1 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1
Bacterial Infection, NOS (Infections and infestations) | 3 | 2
Blood Infection, Bacterial (Infections and infestations) | 1 | 2
Blood Infection, Viral (Infections and infestations) | 1 | 3
Bone Marrow Infection, Viral (Infections and infestations) | 0 | 1
Bradycardic Arrest (Cardiac disorders) | 0 | 1
Brain Infarction (Vascular disorders) | 0 | 1
Cardiac Arrhythmia (Cardiac disorders) | 0 | 1
Chronic Graft vs. Host Disease (General disorders) | 1 | 0
Decreased Consciousness and Delirium (Psychiatric disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 1
Difficulty with Speech (Nervous system disorders) | 0 | 1
Eye Infection, NOS (Infections and infestations) | 0 | 1
Fibrous Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fungal Infection, NOS (Infections and infestations) | 1 | 0
Gastrointestinal Infection, Bacterial (Infections and infestations) | 0 | 1
Gastrointestinal Infection, Fungal (Infections and infestations) | 1 | 0
Genitourinary Hemorrhage (Renal and urinary disorders) | 0 | 1
Genitourinary Infection, Bacterial (Infections and infestations) | 3 | 1
Genitourinary Infection, Fungal (Infections and infestations) | 0 | 1
Genitourinary Infection, Viral (Infections and infestations) | 0 | 1
Graft vs. Host Disease, NOS (General disorders) | 0 | 1
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 | 2
Hemorrhagic Cystitis (Renal and urinary disorders) | 0 | 1
Hypovolemia (Blood and lymphatic system disorders) | 0 | 1
Mucosal Infection, Viral (Infections and infestations) | 1 | 0
Multi-System Organ Failure (General disorders) | 0 | 1
Nervous System Infection, Viral (Infections and infestations) | 1 | 0
Neuropathy (Nervous system disorders) | 0 | 1
New Q Wave (Cardiac disorders) | 0 | 1
Pachymeningeal Thickening (Nervous system disorders) | 0 | 1
Pancreatitis, NOS (Gastrointestinal disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 3 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Requires Dialysis, NOS (Renal and urinary disorders) | 1 | 1
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Infection, Bacterial (Infections and infestations) | 0 | 1
Respiratory Infection, NOS (Infections and infestations) | 1 | 2
Retinal Hemorrhage (Eye disorders) | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Seizures (Nervous system disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Slow Thinking and Movement (Nervous system disorders) | 0 | 1
Small Bowel Obstruction (Gastrointestinal disorders) | 0 | 1
Splenic Infarcts (Vascular disorders) | 0 | 1
Status Epilepticus after Seizures (Nervous system disorders) | 0 | 1
Systolic Ejection Murmur (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Tubular Adenoma, Rectum (Gastrointestinal disorders) | 1 | 0
Viral Infection, NOS (Infections and infestations) | 0 | 3
Wound Infection, Bacterial (Infections and infestations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-10-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT00167180/Prot_SAP_000.pdf